CLINICAL TRIAL: NCT00755222
Title: A Phase 2b, Double-Blind, Randomized, Placebo-Controlled Study of the Safety and Effectiveness of AA4500 Administered Two Times a Week for Up to Three Treatment Cycles (2 x 3) in Subjects With Peyronie's Disease
Brief Title: The Safety and Effectiveness of AA4500 in Subjects With Peyronie's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Endo Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AUX-CC-801
Record Dates: First submitted 2008-09-16; First posted 2008-09-18 (Estimated); Results first posted 2011-04-26 (Estimated); Last update posted 2017-10-05 (Actual); Status verified 2017-09

CONDITIONS: Peyronie's Disease
Keywords: Peyronie's disease; penile plaque; penile curvature
MeSH Terms: conditions — Penile Induration | interventions — Injections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- AA4500 (Experimental): Clostridial collagenase for injection
  Interventions: Biological: AA4500
- Placebo (Placebo Comparator)
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: AA4500 — 2 single injections of study drug per each treatment series up to three treatment series total in study. Each treatment series was separated by 6 weeks.
  Other Names: Clostridial collagenase for injection (AA4500)
  Arms: AA4500
Biological: Placebo — 2 single injections of study drug per each treatment series up to three treatment series total in study. Each treatment series is separated by 6 weeks.
  Arms: Placebo

SUMMARY:
This study evaluated the safety and effectiveness of AA4500 in improving the impact of Peyronie's disease on quality of life and improving penile curvature in men with Peyronie's disease

DETAILED DESCRIPTION:
A Phase 2b randomized, double-blind, placebo-controlled study of AA4500 in the treatment of subjects with Peyronie's disease.

During the screening period, subjects had a physical examination including body weight and height, vital sign measurements, a 12-lead electrocardiogram (ECG), and clinical laboratory testing. Medical history, prior and concomitant medications, and demographic data were recorded.

ELIGIBILITY:
Inclusion Criteria:

* Heterosexual male ≥ 18 years of age
* In a stable relationship with a partner/spouse for at least 3 months before screening
* Have a diagnosis of Peyronie's disease for at least 6 months before first dose of study drug
* Have a penile curvature of at least 30° in the dorsal, lateral, or dorsal/lateral plane
* Have functional difficulty related to Peyronie's disease (eg, difficulty with intromission or erectile dysfunction)
* Be judged to be in good health based upon the results of medical history, physical examination and laboratory profile
* Voluntarily sign an informed consent agreement approved by the Institutional Review Board/Independent Ethics Committee (IRB/IEC). The subject must have also signed an authorization form to allow disclosure of his protected health information. The protected health information authorization form and informed consent form may have been an integrated form or may have been separate forms, depending on the institution
* Be able to complete and understand the various rating instruments

Exclusion Criteria:

* Have had an average of three successive blood pressure readings ≥ 160/100 mmHg during screening or the Day 1 assessments
* Severe pain during penile palpation
* Any of the following conditions:

  * Chordee in the presence or absence of hypospadias
  * Thrombosis of the dorsal penile artery
  * Infiltration by a benign or malignant mass resulting in penile curvature
  * Infiltration by an infectious agent, such as lymphogranuloma venereum
  * Ventral curvature from any cause
  * Presence of sexually transmitted disease
  * Known Hepatitis B or C
  * Known immune deficiency disease or be positive for human immunodeficiency virus (HIV)
* Previously undergone surgery for Peyronie's disease
* Penile curvature of less than 30° or greater than 90°
* Failed to have a rigid erection after pharmacological stimulation with a vasoactive injection of Prostaglandin E1 10 to 20 µg, which, in the opinion of the investigator, was sufficient to accurately measure the subject's penile deformity
* Had a calcified plaque as evident by appropriate radiographic evaluation, penile x-ray, or penile ultrasound. Non-contiguous stippling of calcium was acceptable for inclusion
* Had an isolated hourglass deformity of the penis without curvature
* Had the plaque causing curvature of the penis located proximal to the base of the penis, so that the injection of the local anesthetic would have interfered with the injection of AA4500 into the plaque
* Received alternative medical therapies for Peyronie's disease administered by the intralesional route (including, but not limited to, steroids, verapamil, and the naturally occurring low molecular weight protein, interferon-α2b) within 3 months before the first dose of study drug or plans to use any of these medical therapies at any time during the study
* Received alternative medical therapies for Peyronie's disease administered by the oral (including, but not limited to, vitamin E (>500IU), potassium aminobenzoate [Potaba], tamoxifen, colchicine, pentoxifylline, over-the-counter erectile dysfunction medications, or steroidal anti inflammatory drugs) or topical routes (including, but not limited to, verapamil applied as a cream) within 4 weeks before the first dose of study drug or plans to use any of these medical therapies at any time during the study
* Used any mechanical type device for correction of Peyronie's disease within the 2-week period before screening or plans to use any these devices at any time during the study
* Used a mechanical device to induce a passive erection within the 2-week period before screening or plans to use any of these devices at any time during the study
* Significant erectile dysfunction that has failed to respond to oral treatment with phosphodiesterase type 5 (PDE5) inhibitors
* Recent history of stroke, bleeding, or other medical condition, which in the investigator's opinion would make the subject unsuitable for enrollment in the study
* Unwilling or unable to cooperate with the requirements of the study including completion of all scheduled study visits
* Received an investigational drug or treatment within 30 days before the first dose of study drug
* Allergy to collagenase or any other excipient of AA4500
* Allergy to any concomitant medication required as per the protocol
* Received anticoagulant medication (except for ≤ 165 mg aspirin daily or ≤ 800 mg of over-the-counter NSAIDS daily) during the 7 days before each dose of study drug
* Received doxycycline or a tetracycline derivative during the 7 days before each dose of study drug or plans to use these drugs within 2 days after the injection of study drug
* Received any collagenase treatments within 30 days of the first dose of study drug

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 147 (Actual)
Dates: Start 2008-08; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Veronica Urdaneta, MD, Study Director — Endo Pharmaceuticals
Locations (12):
- United States (12):
  - Urology Associates Medical Group, Burbank, California
  - Urology Specialists Connecticut Clinical Research Center, LLC, Middlebury, Connecticut
  - The Urology Center, PC, New Haven, Connecticut
  - South Florida Medical Research, Aventura, Florida
  - Urology Specialists, SC, Chicago, Illinois
  - Northeast Indiana Research, LLC, Fort Wayne, Indiana
  - Metropolitan Urology, PSC, Jeffersonville, Indiana
  - Maimonides Medical Center Divison of Urology, Brooklyn, New York
  - University Urology Associates, New York, New York
  - Tristate Urologic Services, Cincinnati, Ohio
  - Baylor College of Medicine, Scott Department of Urology, Houston, Texas
  - Urology of Virginia (a division of Sentara Medical Group), Norfolk, Virginia

RESULTS

PARTICIPANT FLOW:
Groups:
- AA4500: Clostridial collagenase for injection 0.58 mg. Study drug was injected directly into the penile plaque (point of maximal concavity as determined by a standard method) of the flaccid penis. Subjects could recieve up to 3 treatment series. During each treatment series, subjects will receive 2 injections of study drug with at least 24 hours but not more than 72 hours between injections.
- Placebo: Placebo was injected directly into the penile plaque (point of maximal concavity as determined by a standard method) of the flaccid penis. Subjects could recieve up to 3 treatment series. During each treatment series, subjects will receive 2 injections of study drug with at least 24 hours but not more than 72 hours between injections.
Period: Overall Study
Arm/Group | AA4500 | Placebo
Started | 111 | 36
Completed | 103 | 34
Not Completed | 8 | 2
Not completed — Withdrawal by Subject | 4 | 2
Not completed — Adverse Event | 2 | 0
Not completed — Protocol Violation | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AA4500 | Placebo | Total
Number analyzed (Participants) | 111 | 36 | 147
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 95 | 34 | 129
  >=65 years | 16 | 2 | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.9 (7.79) | 55.4 (6.95) | 56.6 (7.60)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 111 | 36 | 147
Region of Enrollment [Number; unit: participants]
  United States | 111 | 36 | 147

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Penile Curvature
Description: Negative change reflects improvement in penile curvature
Time Frame: Baseline and Week 36 or last observation carried forward (LOCF)
Measure: Mean (Standard Deviation); unit: Percent change from baseline
Arm/Group | AA4500 | Placebo
Number analyzed (Participants) | 109 | 36
Percent change from baseline | -29.7 (27.16) | -11.0 (30.87)
Statistical Analysis 1: Comparison: AA4500 vs Placebo; Test type: Superiority or Other; p = 0.001, ANOVA

2. Primary Outcome: Change From Baseline in Peyronie's Disease Questionnaire (PDQ) Peyronie's Disease Symptom Bother
Description: Peyronie's disease Symptom Bother Scale: 0-20 lower numbers reflect 'less symptom bother'; higher numbers reflect 'more symptom bother'
  Change from baseline equals Week 36 minus baseline. Negative change reflects improvement in the symptom bother scale.
Time Frame: Baseline to Week 36 or LOCF
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | AA4500 | Placebo
Number analyzed (Participants) | 100 | 34
scores on a scale | -2.6 (4.63) | -0.8 (3.63)
Statistical Analysis 1: Comparison: AA4500 vs Placebo; Test type: Superiority or Other; p = 0.046, ANOVA

3. Primary Outcome: Change From Baseline in PDQ Intercourse Contraint
Description: Peyronie's disease intercourse contraint Scale: 0-12 lower numbers reflect 'less intercourse contraint'; higher numbers reflect 'more intercourse constraint'
  Change from baseline equals Week 36 minus baseline. Negative change reflects improvement in the intercourse constraint scale.
Time Frame: Baseline to Week 36 or LOCF
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | AA4500 | Placebo
Number analyzed (Participants) | 100 | 34
scores on a scale | -1.5 (3.31) | -0.7 (3.65)
Statistical Analysis 1: Comparison: AA4500 vs Placebo; Test type: Superiority or Other; p = 0.164, ANOVA

4. Primary Outcome: Change From Baseline in PDQ Intercourse Discomfort
Description: Peyronie's disease intercourse discomfort Scale: 0-15 lower numbers reflect 'less intercourse discomfort'; higher numbers reflect 'more intercourse discomfort'
  Change from baseline equals Week 36 minus baseline. Negative change reflects improvement in the intercourse discomfort scale.
Time Frame: Baseline to Week 36 or LOCF
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | AA4500 | Placebo
Number analyzed (Participants) | 100 | 34
scores on a scale | -0.8 (3.46) | -0.4 (4.27)
Statistical Analysis 1: Comparison: AA4500 vs Placebo; Test type: Superiority or Other; p = 0.442, ANOVA

5. Primary Outcome: Change From Baseline in PDQ Penile Pain
Description: Peyronie's disease penile pain Scale: 0-40 lower numbers reflect 'less penile pain'; higher numbers reflect 'more penile pain' Change from baseline=Week 36 minus baseline. Negative change reflects improvement in the penile pain scale.
Time Frame: Baseline to Week 36 or LOCF
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | AA4500 | Placebo
Number analyzed (Participants) | 100 | 34
scores on a scale | -2.4 (6.32) | -0.5 (5.30)
Statistical Analysis 1: Comparison: AA4500 vs Placebo; Test type: Superiority or Other; p = 0.095, ANOVA

ADVERSE EVENTS:
Arm/Group | AA4500 | Placebo
Serious Adverse Events (participants affected / at risk) | 4/111 | 1/36
Other Adverse Events (participants affected / at risk) | 109/111 | 28/36
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AA4500 (N=111) | Placebo (N=36)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AA4500 (N=111) | Placebo (N=36)
Injection site bruising (General disorders) | 100 (236) | 18 (36)
Injection site edema (General disorders) | 55 (87) | 0 (0)
Injection site pain (General disorders) | 61 (109) | 5 (7)
Injection site pruritus (General disorders) | 6 (8) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 25 (42) | 2 (4)
General disorder male (Reproductive system and breast disorders) | 6 (7) | 2 (3)
Painful erection (Reproductive system and breast disorders) | 7 (9) | 1 (1)
Penile edema (Reproductive system and breast disorders) | 14 (17) | 1 (1)
Penile pain (Reproductive system and breast disorders) | 14 (14) | 0 (0)
Peyronie's disease (Reproductive system and breast disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Other disclosure agreement that restricts the right of the PI to discuss or publish trial results after the trial is completed.

Auxilium Pharmaceuticals, Inc. agreements may vary with individual investigators but will not prohibit any investigator from publishing. Auxilium supports the publication of results from all centers of a multicenter trial but requests that reports based on single site data not preceed the primary publication of the entire clinical trial.